CLINICAL TRIAL: NCT05786001
Title: Evaluation of Lower Limb Angiosome Perfusion and Oxygenation Using Thermal and Hyperspectral Imaging
Brief Title: Multimodal Noninvasive Assessment of Peripheral Circulation in Chronic Limb-threatening Ischemia
Status: Recruiting | Type: Observational
Sponsor: Tampere University (Other)
Collaborators: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Niku Oksala, Prof, MD, PhD, DSc, Tampere University
Other Study IDs: R20156L
Record Dates: First submitted 2023-01-30; First posted 2023-03-27 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Chronic Limb Threatening Ischemia
Keywords: hyperspectral imaging; thermal imaging; angiosomes; CLTI; diabetes
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (3):
- Unhealthy group: Individuals with CLTI
- Age control group: Healthy individuals over the age of 50
- Healthy group: Healthy and young individuals

SUMMARY:
Assessment of a novel diagnostic method for screening and diagnosing chronic limb-threatening ischemia (CLTI). Using hyperspectral and thermal imaging, the perfusion and oxygenation in the lower limbs will be studied in healthy and unhealthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* for CLTI patients age >50
* for age control group age >50 and not diagnosed with cardiovascular diseases. 0.9 < ABI < 1.3
* for healthy group 18 <= age <= 50 and no history of cardiovascular disease
* volunteering for study

Exclusion Criteria:

* inability to give informed consent
* denial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * patients at the Vascular Centre Polyclinic and Vascular Surgery Ward at Tampere University Hospital
  * Orthopaedic patients, joint replacement hospital and orthopaedic ward at Tampere University Hospital
  * students and staff from Tampere University and Tampere University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Perfusion in lower limb angiosomes assessed by thermal imaging | 45 minutes during the procedure starting from the first measurement and ending after the last measurement
  Thermal imaging will be used to assess the perfusion in the lower limbs. The lower limb can be divided into six angiosomes, which can then be used to assess thermal patterns. Healthy and unhealthy feet will present with different thermal patterns and other changes in thermographs.
Oxygenation in lower limb angiosomes assessed by hyperspectral imaging. | 45 minutes during the procedure starting from the first measurement and ending after the last measurement
  Hyperspectral imaging can be used in the assessment of oxygenation in the lower limb angiosomes. Based on hyperspectral imaging, oxygenation maps can be generated and then analyzed. Differences between the oxygenation maps of healthy and unhealthy patients will be established.

CONTACTS AND LOCATIONS:
Overall Officials: Niku Oksala, MD, PhD, DSc, Principal Investigator — Tampere University, Tampere University Hospital
Locations (1):
- Tampere University, Tampere, Pirkanmaa, Finland